CLINICAL TRIAL: NCT01654367
Title: The Effectiveness and Safety of Treating Operable Breast Cancer by the Adjuvant Therapy of Zoledronic Acid and Aromatase Inhibitors and/or Ovarian Function Inhibition
Brief Title: Research of Zoledronic Acid and Aromatase Inhibitors as Adjuvant Therapy to Breast Cancer
Acronym: esozao
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Zhang jin, Tianjin Medical University, Tianjin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jzhang2
Record Dates: First submitted 2012-07-19; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zoledronic Acid and Aromatase Inhibitors (Experimental): Zoledronic Acid and Aromatase Inhibitors for Adjuvant Therapy
  Interventions: Drug: Zoledronic Acid and Aromatase Inhibitors

INTERVENTIONS:
Drug: Zoledronic Acid and Aromatase Inhibitors — Zoledronic Acid and Aromatase Inhibitors as Adjuvant Therapy

SUMMARY:
Select patients of primary breast cancer whose hormone receptor is positive and accepted postoperative adjuvant aromatase inhibitors for endocrine treatment.Treat them with zoledronic acid 4mg intravenous infusion every six months until the end of the aromatase treatment. Assess the disease-free survival; overall survival; combination of security, as well as the situation of bone loss.

DETAILED DESCRIPTION:
The investigators select patients of primary breast cancer whose hormone receptor is positive and accepted postoperative adjuvant aromatase inhibitors for endocrine treatment.Treat them with zoledronic acid 4mg intravenous infusion every six months until the end of the aromatase treatment. Assess the disease-free survival; overall survival; combination of security, as well as the situation of bone loss.

ELIGIBILITY:
Inclusion Criteria:

1. Karnofsky≥70
2. Provision of informed consent
3. Pathological confirmation of breast cancer
4. Hormone receptor-positive and accept aromatase inhibitors for adjuvant endocrine therapy
5. Not previously received treatment with bisphosphonate
6. Laboratory criteria:

   PLT≥100*109/L WBC≥4000/mm3 HGB≥10g/dl GOT,GPT,ALP≤2*ULN TBIL,DBIL,CCr≤1.5*ULN
7. Surgery , radiotherapy and chemotherapy has finished

Exclusion Criteria:

1. Pregnant of lactation woman
2. History of organ transplantation
3. With mental disease
4. With severe infection or active gastrointestinal ulcers
5. With severe liver disease (such as cirrhosis), kidney disease, respiratory disease or diabetes
6. Disease-free period of other malignant tumor is less than 5 years(except cured basal cell skin cancer and cervical carcinoma in situ)
7. With heart disease
8. Experimental drug allergy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
therapeutic assessment | 6 months
  therapeutic assessment

SECONDARY OUTCOMES:
Adverse reactions and disease-free survival | 2 years
  Adverse reactions and disease-free survival

OTHER OUTCOMES:
Recurrence or death | 5 years
  Recurrence or death

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhang, Professor, Study Chair — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China